CLINICAL TRIAL: NCT00782275
Title: A Phase II Trial of Avastin and Temsirolimus Following Tyrosine Kinase Inhibitor Failure in Patients With Advanced Renal Cell Carcinoma
Brief Title: Avastin and Temsirolimus Following Tyrosine Kinase Inhibitor Failure in Patients With Advanced Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Genentech, Inc. (Industry); Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David F. McDermott, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-184
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Results first posted 2017-12-20 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Renal Cell Carcinoma; Kidney Cancer
Keywords: RCC; avastin; temsirolimus
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Bevacizumab; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bevacizumab and temsirolimus (Experimental): bevacizumab: given intravenously at a dose of 10mg/kg every 2 weeks (days 1 and 15)
  temsirolimus: given intravenously at a dose of 25mg weekly on days 1, 8, 15, and 22
  1 cycle=28-days
  There were no dose reductions for bevacizumab allowed. If bevacizumab was held, the same dose would be used if treatment were resumed. If temsirolimus was held, the same or a reduced dose (15mg IV weekly) could be used upon resumption of therapy. Treatment was continued until the development of unacceptable toxicity or progression.
  Interventions: Drug: bevacizumab; Drug: temsirolimus

INTERVENTIONS:
Drug: bevacizumab
  Other Names: avastin
Drug: temsirolimus
  Other Names: torisel

SUMMARY:
This is a single-arm phase II trial evaluating the combination of avastin and temsirolimus in patients with metastatic renal cell cancer (RCC) including both histologically confirmed clear cell (cc) or non-clear cell (ncc) subtypes. Patients must have experienced disease progression or intolerable toxicity with a vascular endothelial growth factor (VEGF)-targeted tyrosine kinase inhibitor (TKI) (e.g. sorafenib, sunitinib, pazopanib). Only 2 prior VEGF therapies are allowed. The purpose of this research study is to evaluate efficacy of the combination against an historical control. Temsirolimus has been approved by the Food and Drug Administration (FDA) in the treatment of renal cell carcinoma. Avastin has been approved by the FDA for other types of cancers but not renal cell carcinoma.

DETAILED DESCRIPTION:
Avastin, a humanized IgG1 monoclonal antibody (MAb), inhibits vascular endothelial growth factor (VEGF). VEGF is one of the most potent and specific proangiogenic factors and has been identified as a crucial regulator of both normal and pathological angiogenesis. Temsirolimus specifically inhibits the mammalian target of rapamycin (mTOR), a highly conserved serine/threonine kinase which regulates cell growth and metabolism in response to environmental factors. The combination avastin and temsirolimus has already demonstrated efficacy in the phase I setting

STATISTICAL CONSIDERATIONS:

The primary endpoint is 4-month PFS. The null and alternative hypotheses are 50% vs. 70%. Assuming 2 ineligible patients, the target sample size is 41 patients (39 eligible patients). The probability of concluding that the treatment is effective was >0.90 if the true rate is at least 70%. The probability of concluding that the treatment is effective was ≤ 0.10 if the true rate was 50% or less. If 24 or more patients are alive and progression-free at 4 months, then this regimen would be considered for further study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed renal cell carcinoma in either primary or metastatic lesions. Non-clear histology will be allowed.
* Disease progression on a VEGF-targeted tyrosine kinase inhibitor as the most recent therapy or have experienced intolerable toxicity so as require discontinuation. Only one prior VEGF-targeted tyrosine kinase inhibitor.
* Must be off of VEGF-targeted tyrosine kinase inhibitor for 2 weeks or greater.
* One measurable lesion which is not curable by standard radiation therapy or surgery.
* The enrolling site must agree to obtain paraffin-embedded tumor blocks or at least 10 unstained, paraffin-embedded slides for submission for correlative studies.
* 18 years of age or older
* ECOG Performance Status of 0 or 1
* Baseline laboratory values as outlined in the protocol
* Life expectancy of greater than 3 months
* No prior malignancy diagnosed within the past three years, other than superficial basal cell and superficial squamous cell, or carcinoma in situ of the cervix.

Exclusion Criteria:

* Known CNS disease, except for treated brain metastases
* Previously treated with avastin or mTOR inhibitors
* Other then VEFG-targeted TKI, patients may only have had prior immunotherapy or chemotherapy for stage IV disease
* History of allergic reaction to Chinese hamster ovary cell products, other recombinant antibodies, or compounds of similar chemical or biologic composition to avastin or temsirolimus
* History of bleeding diathesis or coagulopathy. Therapeutic anticoagulants are allowed
* Patients with clinically significant cardiovascular disease
* Patients receiving enzyme-inducing antiepileptic drugs or any other CYP3A4 inducer such as rifampin or St. John's wort
* No serious non-healing wound, ulcer or bone fracture
* No uncontrolled intercurrent illness including , but not limited to, ongoing active infection requiring parental antibiotics or psychiatric illness/social situations that would limit compliance with study requirements
* HIV-positive receiving combination anti-retroviral therapy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of vascular access device, within 7 days prior to enrollment on study
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Known hypersensitivity to any component of avastin or temsirolimus
* Life expectancy of less than 12 weeks
* History of hemoptysis within 1 month prior to day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David McDermott, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Vanderbilt Univeristy Medical Center, Nashville, Tennessee

REFERENCES:
- [Result] Mahoney KM, Jacobus S, Bhatt RS, Song J, Carvo I, Cheng SC, Simpson M, Fay AP, Puzanov I, Michaelson MD, Atkins MB, McDermott DF, Signoretti S, Choueiri TK. Phase 2 Study of Bevacizumab and Temsirolimus After VEGFR TKI in Metastatic Renal Cell Carcinoma. Clin Genitourin Cancer. 2016 Aug;14(4):304-313.e6. doi: 10.1016/j.clgc.2016.02.007. Epub 2016 Feb 23. PMID 27036973

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between April 2009 and May 2013.
Groups:
- Bevacizumab + Temsirolimus: bevacizumab: given intravenously at a dose of 10mg/kg every 2 weeks (days 1 and 15)
  temsirolimus: given intravenously at a dose of 25mg weekly on days 1, 8, 15, and 22
  1 cycle=28 days
  There were no dose reductions for bevacizumab allowed. If bevacizumab was held, the same dose would be used if treatment were resumed. If temsirolimus was held, the same or a reduced dose (15mg IV weekly) could be used upon resumption of therapy. Treatment was continued until the development of unacceptable toxicity or progression.
Period: Overall Study
Arm/Group | Bevacizumab + Temsirolimus
Started | 41
Treated | 40
Prior VEGFR Response Evaluable (Pts were classified by response to previous VEGFR TKI therapy at baseline: refractory or responsive.) | 39 (One patient was unevaluable and therefore excluded from related subgroup analyses.)
Completed | 0 (Since treatment duration was not fixed, patients were not considered to have completed treatment.)
Not Completed | 41
Not completed — Adverse Event | 11
Not completed — Withdrawal by Subject | 1
Not completed — Progressive Disease | 21
Not completed — Physician Decision | 4
Not completed — Not started treatment | 1
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all treated patients as opposed to enrolled patients.
Arm/Group | Bevacizumab + Temsirolimus
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 60 [32 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 33
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40
Primary VEGF Refractory Status [Count of Participants; unit: Participants] — Primary VEGF refractory status was based on the prior therapy form; patients were considered refractory if response on prior therapy was progressive disease OR prior therapy duration was < 3 months and patient experienced progression at the end of therapy. Population: One patient did not have enough data to determine VEGF-refractory status.
  Participants
    VEGF Refractory-No | 20
    VEGF Refractory-Yes | 19
    Unevaluable | 1
MSKCC Risk Category [Count of Participants; unit: Participants] — The Memorial Sloan Kettering Cancer Center (MSKCC) risk score is based on the sum of positive answers to the following criteria: 1) time from the earliest of initial or metastatic diagnosis to first prior treatment < 1 year; 2) Karnofsky Performance Score < 80%; 3) HgB < LLN; 4) Corrected Calcium > 10 mg/dL; and 5) NLDH> 1.5xULN. Patients were further classified into risk groups based on the score of 0=Favorable, 1-2=Intermediate and 3-5=Poor Risk. (Motzer et al. Cancer 2008; 113)
  Participants
    Favorable | 5
    Intermediate | 31
    Poor | 4

OUTCOME MEASURES:

1. Primary Outcome: 4-month Progression-Free Survival Rate
Description: 4-month progression-free survival rate was defined as the percentage of participants absent death or progression based on Response Evaluation Criteria In Solid Tumors Criteria (RECIST) before 4 months. Per RECIST 1.0 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease evaluations occurred every 8 weeks (+/- 1 wk) on treatment. Relevant for this endpoint was disease status at 4 months.
Population: The analysis dataset is comprised of all treated participants.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Temsirolimus
Number analyzed (Participants) | 40
percentage of participants | 65 [50.8 to 77.5]
Statistical Analysis 1: Comparison: Bevacizumab + Temsirolimus; The regimen was evaluated against an historical control with null and alternative 4-month PFS rates of 50% and 70%, respectively. With the final sample size of 40 eligible patients and using the same operating characteristics (alpha and beta 10%), the decision rule changes such that if 25 or more patients of 40 are alive and progression-free at 4 months then this regimen is considered promising; Test type: Superiority; p = 0.081, exact binomial test

2. Secondary Outcome: Objective Response Rate
Description: Objective response (OR) rate is the percentage of participants achieving partial response (PR) or complete response (CR) based on RECIST 1.0 criteria on treatment. Per RECIST 1.0 for target lesions, CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. To be assigned a status of CR or PR, changes in tumor measurements must be confirmed by repeat assessments performed no fewer than 4 weeks after the response criteria are first met. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Disease evaluations occurred every 8 weeks (+/- 1 wk) on treatment; Treatment continued until disease progression or unacceptable toxicity. Median (range) of treatment duration for this study cohort was 5 cycles (1-39) [1 cycle=28days].
Population: The analysis dataset is comprised of all treated participants.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Temsirolimus
Number analyzed (Participants) | 40
percentage of participants | 17.5 [8.5 to 30.4]

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined from the date of registration to date of death, or censored at the date the participant was last known alive. OS is estimated based on the Kaplan-Meier method.
Time Frame: Median follow-up for survival in this study cohort is 56 months.
Population: The analysis dataset is comprised of all treated participants.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Temsirolimus
Number analyzed (Participants) | 40
months | 12.2 [7.7 to 21.9]

ADVERSE EVENTS:
Time Frame: Assessed each cycle throughout treatment from time of first dose and up to day 30 post-treatment. Treatment duration in cycles was a median (range) of 5 (1-39) which parallels time in months given the 28 day cycle duration.
Description: Maximum grade toxicity by type was first calculated including events only with temsirolimus and/or bevacizumab treatment-attribution of possibly, probably or definitely. Serious AEs were defined as grade 3 or higher events per CTCAEv3. Other AEs were defined as grades 1 or 2 events per CTCAEv3. No further data is available to specify classification of 'other' beyond the general term.
Arm/Group | Bevacizumab + Temsirolimus
Serious Adverse Events (participants affected / at risk) | 28/40
Other Adverse Events (participants affected / at risk) | 38/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Temsirolimus (N=40)
Hemoglobin (Blood and lymphatic system disorders) | 2
Ventricular arrhythmia NOS (Cardiac disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Fistula, Esophageal (Gastrointestinal disorders) | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 1
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Lower GI, hemorrhage NOS (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 4
Fever w/o neutropenia (General disorders) | 1
Edema limb (General disorders) | 1
Syndromes-other (General disorders) | 1
Infection w/ unk ANC skin (cellulitis) (Infections and infestations) | 1
Infection w/ unk ANC blood (Infections and infestations) | 1
Wound - non-infectious (Injury, poisoning and procedural complications) | 1
Vascular access,Thrombosis/embolism (Injury, poisoning and procedural complications) | 1
Haptoglobin (Investigations) | 1
Neutrophils (Investigations) | 1
Weight gain (Investigations) | 1
PTT (Investigations) | 1
Alkaline phosphatase (Investigations) | 1
ALT, SGPT (Investigations) | 1
AST, SGOT (Investigations) | 2
Hypercholesterolemia (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 6
Neck, pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Head/headache (Nervous system disorders) | 1
Glomerular filtration rate (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 4
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 5
Hypotension (Vascular disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1
Pulmonary/ Upper Respiratory- other (Respiratory, thoracic and mediastinal disorders) | 1
Rash/ desquamation (Skin and subcutaneous tissue disorders) | 1
Thrombosis/ thrombus/ embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Temsirolimus (N=40)
Hemorrhage-other (Blood and lymphatic system disorders) | 1
Hemoglobinuria (Blood and lymphatic system disorders) | 2
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 13
Hematologic-other (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Arrhythmia-other (Cardiac disorders) | 1
Cardiac-other (Cardiac disorders) | 1
Tearing (Eye disorders) | 1
Ocular-other (Eye disorders) | 3
Eye, pain (Eye disorders) | 1
Chelitis (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Periodontal disease (Gastrointestinal disorders) | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 10
Distention/bloating, abdominal (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 3
Hemorrhoids (Gastrointestinal disorders) | 2
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 10
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 8
GI-other (Gastrointestinal disorders) | 8
Oral cavity, hemorrhage (Gastrointestinal disorders) | 2
Rectum, hemorrhage (Gastrointestinal disorders) | 1
Abdomen, pain (Gastrointestinal disorders) | 3
Anus, pain (Gastrointestinal disorders) | 1
Dental/teeth/peridontal, pain (Gastrointestinal disorders) | 1
Oral cavity, pain (Gastrointestinal disorders) | 1
Oral gums, pain (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 20
Fever w/o neutropenia (General disorders) | 4
Rigors/chills (General disorders) | 2
Constitutional, other (General disorders) | 4
Edema head and neck (General disorders) | 1
Edema limb (General disorders) | 7
Edema trunk/genital (General disorders) | 1
Chest/thoracic pain NOS (General disorders) | 2
Face, pain (General disorders) | 1
Pain-other (General disorders) | 5
Allergy-other (Immune system disorders) | 3
Infection Gr0-2 neut, sinus (Infections and infestations) | 2
Infection Gr0-2 neut, skin (Infections and infestations) | 1
Infection w/ unk ANC nerve-peripheral (Infections and infestations) | 1
Infection-other (Infections and infestations) | 4
Bruising (Injury, poisoning and procedural complications) | 3
Leukocytes (Investigations) | 3
Lymphopenia (Investigations) | 5
Platelets (Investigations) | 4
Weight gain (Investigations) | 1
Weight loss (Investigations) | 12
INR (Investigations) | 3
PTT (Investigations) | 3
Alkaline phosphatase (Investigations) | 2
ALT, SGPT (Investigations) | 6
AST, SGOT (Investigations) | 7
Hypercholesterolemia (Investigations) | 15
Creatinine (Investigations) | 11
Metabolic/Laboratory-other (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 14
Dehydration (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 14
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 1
Back, pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 2
Joint, pain (Musculoskeletal and connective tissue disorders) | 4
Muscle, pain (Musculoskeletal and connective tissue disorders) | 1
Taste disturbance (Nervous system disorders) | 6
Dizziness (Nervous system disorders) | 1
Neuropathy-motor (Nervous system disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 2
Neurologic-other (Nervous system disorders) | 1
Head/headache (Nervous system disorders) | 10
Sinus, pain (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 2
Urinary hemorrhage NOS (Renal and urinary disorders) | 2
Glomerular filtration rate (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 12
Renal/GU-other (Renal and urinary disorders) | 1
Erectile impotence (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Muco/stomatitis (symptom) larynx (Respiratory, thoracic and mediastinal disorders) | 1
Muco/stomatitis (symptom) pharynx (Respiratory, thoracic and mediastinal disorders) | 1
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 15
Pleura, pain (Respiratory, thoracic and mediastinal disorders) | 1
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 9
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 7
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 9
Sweating (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 8
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 2
Pruritus/itching (Skin and subcutaneous tissue disorders) | 12
Rash/desquamation (Skin and subcutaneous tissue disorders) | 9
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 12
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 6
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Skin-other (Skin and subcutaneous tissue disorders) | 7
Scalp, pain (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Hemorrhage-other (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No